CLINICAL TRIAL: NCT03221309
Title: A Novel Model of Hepatitis C Treatment as Anchor to Prevent HIV, Initiate Opioid Substitution Therapy, and Reduce Risky Behavior
Brief Title: Hepatitis C Treatment to Prevent HIV, Initiate Opioid Substitution Therapy, and Reduce Risky Behavior
Acronym: ANCHOR
Status: Active, not recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Elana Rosenthal, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00071577
Record Dates: First submitted 2017-07-13; First posted 2017-07-18 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: HCV; Buprenorphine; PreP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Adults infected with HCV: Phase 1 (first 100 enrolled participants) HCV-infected adults with on-going injection drug use use with opioids with 3 months of screening
  Phase 2 (enrolled participants 101-200) HCV-infected adults with on-going opioid misuse of non-prescription opioids within twelve months of screening
  Interventions: Other: Evaluate model of care for HCV-infected adults with on-going opioid misuse

INTERVENTIONS:
Other: Evaluate model of care for HCV-infected adults with on-going opioid misuse — Participants will be treated with direct-acting antivirals per standard of care and will be concomittantly be offered PreP for HIV prevention and buprenorphine for treatment of opioid-use disorder when clinically indicated

SUMMARY:
This is an open label, non-randomized, observational pilot study to evaluate a model of care for treatment of hepatitis C in people with ongoing injection drug use. Participants will be treated with direct-acting antivirals (DAA) as per standard of care and will concomittantly be offered pre-exposure prophylaxis for HIV prevention and buprenorphine for treatment of opioid use disorder when clinically indicated.

DETAILED DESCRIPTION:
Hepatitis C (HCV) is a chronic infection with significant morbidity and mortality. The development of directly acting antivirals (DAA) has dramatically improved the cure rate of HCV treatment. However, despite the availability of effective therapy, the global epidemic of HCV infection continues to be driven by people with ongoing injection drug use (PWID), who are largely excluded from HCV therapy. Several critical barriers exist preventing high-risk patients' entry to care, including (1) lack of engagement in the traditional healthcare system by marginalized patient populations, and (2) insurance restrictions due to concerns regarding treatment adherence and HCV reinfection. Furthermore, ongoing injection drug use places these individuals at high risk of HIV acquisition. However, studies have repeatedly demonstrated that pre-exposure prophylaxis (PrEP) reduces HIV acquisition and opioid substitution therapy with buprenorphine reduces HIV and HCV acquisition in PWID.

As such, we propose a comprehensive model of care to engage individuals with ongoing injection drug use in treatment of HCV, in conjunction with collocated services to prevent HIV acquisition and HCV reinfection, including pre-exposure prophylaxis and opioid substitution therapy. This pilot trial will demonstrate whether a comprehensive model of care can simultaneously treat HCV, and prevent HCV reinfection, HIV acquisition and effectively treat opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old
2. Able and willing to sign informed consent
3. Chronically infected with HCV, defined as any individual with documentation of positive HCV antibody and positive HCV RNA test (HCV RNA of 2,000 IU/mL or greater).
4. Willing to have samples stored for future use
5. Ongoing injection drug use, defined as self-report of either:

   1. Phase 1 (first 100 enrolled participants) Injection non-prescription drug use within three months of screening visit or
   2. Phase 2 (enrolled participants 101-200) Use of non-prescription opioids within twelve months of screening visit

Exclusion Criteria:

1. Decompensated liver disease (Childs Pugh B or C)
2. Unable to comply with research study visits
3. Poor venous access not allowing screening laboratory collection
4. Have any condition that the investigator considers a contraindication to study participation
5. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults infected with HCV and have on-going misuse with opioids
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elana Rosenthal, MD, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - HIPS, Washington D.C., District of Columbia
  - University of Maryland Drug Treatment Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenthal ES, Silk R, Mathur P, Gross C, Eyasu R, Nussdorf L, Hill K, Brokus C, D'Amore A, Sidique N, Bijole P, Jones M, Kier R, McCullough D, Sternberg D, Stafford K, Sun J, Masur H, Kottilil S, Kattakuzhy S. Concurrent Initiation of Hepatitis C and Opioid Use Disorder Treatment in People Who Inject Drugs. Clin Infect Dis. 2020 Oct 23;71(7):1715-1722. doi: 10.1093/cid/ciaa105. PMID 32009165

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults Infected With HCV: Phase 1 (first 100 enrolled participants) HCV-infected adults with on-going injection drug use use with opioids with 3 months of screening
  Phase 2 (enrolled participants 101-198) HCV-infected adults with on-going opioid misuse of non-prescription opioids within twelve months of screening
  Evaluate model of care for HCV-infected adults with on-going opioid misuse: Participants will be treated with direct-acting antivirals per standard of care and will be concomittantly be offered PreP for HIV prevention and buprenorphine for treatment of opioid-use disorder when clinically indicated
Period: Overall Study
Arm/Group | Adults Infected With HCV
Started | 198
Phase 1 | 100
Phase 2 | 98
Completed | 160
Not Completed | 38

BASELINE CHARACTERISTICS:
Groups:
- Adults Infected With HCV: Phase 1 (first 100 enrolled participants) HCV-infected adults with on-going injection drug use use with opioids with 3 months of screening
  Phase 2 (enrolled participants 101-200) HCV-infected adults with on-going opioid misuse of non-prescription opioids within twelve months of screening
  Evaluate model of care for HCV-infected adults with on-going opioid misuse: Participants will be treated with direct-acting antivirals per standard of care and will be concomittantly be offered PreP for HIV prevention and buprenorphine for treatment of opioid-use disorder when clinically indicated
Arm/Group | Adults Infected With HCV
Number analyzed (Participants) | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 182
  >=65 years | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [52 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 197
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 165
  White | 26
  More than one race | 4
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 198
Chronic HCV Infection [Count of Participants; unit: Participants] | 198

OUTCOME MEASURES:

1. Primary Outcome: Hepatitis C Virus (HCV) Cure (Sustained Virologic Response)
Description: Undetectable HCV viral load 12 weeks after the end of treatment
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Adults Infected With Hepatitis C Virus (HCV): Two Phases:
  Phase 1 (first 100 enrolled participants) HCV-infected adults with on-going injection drug use use with opioids with 3 months of screening
  Phase 2 (enrolled participants 101-198) HCV-infected adults with on-going opioid misuse of non-prescription opioids within twelve months of screening
  Evaluate model of care for HCV-infected adults with on-going opioid misuse: Participants will be treated with direct-acting antivirals per standard of care and will be concomittantly be offered Pre-Exposure Prophylaxis (PrEP) for HIV prevention and buprenorphine for treatment of opioid-use disorder when clinically indicated
Arm/Group | Adults Infected With Hepatitis C Virus (HCV)
Number analyzed (Participants) | 198
Participants | 158

2. Secondary Outcome: Uptake of HIV Pre-exposure Prophylaxis (PrEP)
Description: Number of participants who initiated PrEP between Day 0 and Week 24
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- HIV Negative Adults: 185 HIV negative adults enrolled in ANCHOR study
Arm/Group | HIV Negative Adults
Number analyzed (Participants) | 185
Participants | 29

3. Secondary Outcome: Retention on HIV PrEP
Description: Number of participants who initiated PrEP between Day 0 and Week 24 and continued on PrEP through week 48
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- HIV Negative Adults Who Initiated PrEP: 29 HIV negative adults enrolled in ANCHOR who initiated PrEP between Day 0 and Week 24
Arm/Group | HIV Negative Adults Who Initiated PrEP
Number analyzed (Participants) | 29
Participants | 8

4. Secondary Outcome: Uptake of Buprenorphine
Description: Number of participants who initiated on-site co-located buprenorphine between Day 0 and Week 24
Time Frame: 24 weeks
Population: Patients not on MOUD at time of ANCHOR screening
Measure: Count of Participants; unit: Participants
Groups:
- Adults Not on Medication for Opioid Use Disorder (MOUD): 90 adults with opioid use disorder not on MOUD at ANCHOR screening
Arm/Group | Adults Not on Medication for Opioid Use Disorder (MOUD)
Number analyzed (Participants) | 90
Participants | 61

5. Secondary Outcome: Retention in Buprenorphine Program
Description: Number of participants who initiated buprenorphine between Day 0 and Week 24 and were retained in buprenorphine treatment at week 48
Time Frame: 48 weeks
Population: Patients who initiated buprenorphine between Day 0 and Week 24
Measure: Count of Participants; unit: Participants
Groups:
- Adults Who Initiated Buprenorphine: 61 adults with opioid use disorder who initiated on-site co-located buprenorphine treatment between ANCHOR screening and week 24
Arm/Group | Adults Who Initiated Buprenorphine
Number analyzed (Participants) | 61
Participants | 41

ADVERSE EVENTS:
Time Frame: Through study completion (96 weeks)
Arm/Group | Adults Infected With HCV
All-Cause Mortality (participants affected / at risk) | 14/198
Serious Adverse Events (participants affected / at risk) | 0/198
Other Adverse Events (participants affected / at risk) | 0/198

LIMITATIONS AND CAVEATS:
Study conducted at two urban sites, may not be generalizable to all populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT03221309/Prot_SAP_000.pdf